CLINICAL TRIAL: NCT01872065
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalating Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ARC-520 in Normal Adult Volunteers
Brief Title: Safety and Tolerability Study of ARC-520 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Heparc-1001
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — ARC-520

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ARC-520 (Experimental): Single dose, intravenous administration of ARC-520.
  Interventions: Drug: ARC-520
- Normal Saline (Placebo Comparator): Single dose, intravenous administration of Normal Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARC-520
  Arms: ARC-520
Drug: Placebo
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of ARC-520 in normal, adult volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male or female subjects, 18-55 years of age
* Be a non-smoker

Key Exclusion Criteria:

* History of clinically relevant medical illnesses that in the Investigator opinion may jeopardize subject safety or interfere with participation in the study, including but not limited to hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Acute signs of hepatitis/other infection (e.g., moderate fever, jaundice, nausea, vomiting, abdominal pain) evident within 4 weeks of screening and/or at the screening examination.
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to administration of study treatment.
* Is sero-positive for HIV, HBV, HCV, and/or a history of delta virus hepatitis.
* Currently uses and/or has a history of alcohol and/or drug abuse < 12 months from screening.
* Use of investigational agents or devices within 30 days prior to planned study dosing or current participation in an investigational study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To determine the incidence and frequency of adverse events as a measure of safety and tolerability of ARC-520 | One month
  The incidence and frequency of adverse events (AEs), serious adverse events (SAEs), related AEs, related SAEs, and AEs leading to withdrawal, dose modification, or treatment discontinuation will be summarized by dose and treatment group.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of ARC-520 at different dose concentrations | 2 days
  Plasma concentrations following a single dose of ARC-520 at different dose levels will be used to calculate the following ARC-520 pharmacokinetic parameters: Cmax, tmax, AUC0-24, AUCinf, and t1/2. Descriptive statistics of pharmacokinetic parameters will include mean, standard deviation, and coefficient of variation.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, PhD, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Research Site 1, Melbourne, Victoria, Australia